CLINICAL TRIAL: NCT07153458
Title: Identification of New Non-invasive, Predictive, and Diagnostic Biomarkers for Colorectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis (Other)
Collaborators: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Pasqua Letizia Pesole, Principal Investigator, Azienda Ospedaliera Specializzata in Gastroenterologia Saverio de Bellis
Other Study IDs: RC2025-26; RC2025-26 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2025-08-05; First posted 2025-09-04 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: CRC (Colorectal Cancer); Adenoma Colon
Keywords: crc (colorectal cancer); Adenoma colon; Biomarkers; neoplasm
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients undergoing surgery at the Department of Surgery, with a diagnosis of CRC;: Patients undergoing surgery at the Department of Surgery, with a diagnosis of CRC;
- Subjects with a negative endoscopic examination result.: Subjects who attend our Institution's Department of Digestive Endoscopy for a colonoscopy performed for diagnostic purposes, with a negative endoscopic examination result.
- Subjects with a diagnosis of adenoma with high-grade dysplasia, a condition considered pre-cancerous: Subjects who attend our Institution's Department of Digestive Endoscopy for a colonoscopy performed for diagnostic purposes, or patients undergoing a surgical procedure at the Department of Surgery, in whom the presence of an adenoma with high-grade dysplasia is found, a condition considered pre-cancerous.

SUMMARY:
The study in question is an observational study that aims to identify new non-invasive biomarkers present in the serum of patients with CRC and, subsequently, to create a score capable of predicting the development of CRC.

It is an observational study with 3 enrollment arms:

Arm 1: Patients undergoing surgery at the U.O.C. of Surgery, with a CRC diagnosis;

Arm 2: Subjects with a negative result from the endoscopic examination;

Arm 3: Subjects in whom the presence of an adenoma with high-grade dysplasia is found, a condition considered pre-cancerous.

DETAILED DESCRIPTION:
Given the observational nature of the study, patients who access our Institute for diagnostic tests or procedures planned as part of normal clinical practice will be enrolled.

This study involves three enrollment arms:

Arm 1: Patients undergoing surgery at the Department of Surgery with a diagnosis of CRC;

Arm 2: Subjects who attend our Institution's Department of Digestive Endoscopy for a colonoscopy performed for diagnostic purposes, with a negative endoscopic examination result;

Arm 3: Subjects who attend our Institution's Department of Digestive Endoscopy for a colonoscopy performed for diagnostic purposes, or patients undergoing surgery at the Department of Surgery, in whom the presence of an adenoma with high-grade dysplasia, a condition considered pre-cancerous, will be found.

Patients recruited in Arm 1, should they decide to participate in the study, will sign the prepared informed consent form. They will undergo a family, pathological, and pharmacological history review, and subsequently, a blood sample will be taken. At the follow-up visit, patients will undergo another blood draw. After the surgical procedure, 'leftover tissue' samples-that is, portions of tissue no longer needed for diagnostic purposes-will be collected for the identification of macromolecules (nucleic acids, proteins, carbohydrates, fats, etc.).

Subjects potentially eligible for enrollment in arms 2 and 3, should they decide to participate in the study, will sign the study-specific informed consent form, will undergo a history review, and a subsequent blood sample will be taken.

At the end of the colonoscopy, subjects who are found to be free of disease will be enrolled in Arm 2 and will form the healthy subject cohort. In the event that a suspicious polyp is found during the colonoscopy and a biopsy is taken, the result of the histological examination will be awaited. In the case of a diagnosis of Adenoma with high-grade dysplasia, the subject will be enrolled in Arm 3.

Blood samples taken from subjects enrolled in all study arms will be used for the determination of tumor markers used in clinical practice, such as CEA, CA19.9, and AFP. Any remaining blood samples will be processed to obtain serum and plasma and will be stored in a Biobank. Subsequently, they will be used for the measurement of potential biomarkers, such as FGF-21, PPY, and SOD3, using ELISA (Enzyme-linked Immunosorbent Assay).

Using ATR-FTIR technology (Attenuated Total Reflectance - Fourier Transform Infrared Spectroscopy), serum, plasma, and tissues will be analyzed to determine their composition in terms of macromolecules (nucleic acids, proteins, carbohydrates, fats). The purpose of this investigation will therefore be to identify any alterations in the characteristic absorption profile of the disease. The ATR-FTIR technique is a variant of traditional Fourier Transform Infrared Spectroscopy. In the ATR-FTIR system, broad-spectrum radiation in the IR region is channeled into a Fourier transform spectrometer where the light is made to interfere. Leaving the spectrometer, and before the radiation detector, the radiation is passed through a crystal with a high refractive index, on which the sample to be analyzed is placed. When the light meets the contact surface between the crystal and the sample, it is completely reflected, but an evanescent wave is generated which penetrates the sample to distances on the order of a micrometer. This interaction between the evanescent wave and the sample leads to the selective absorption of the characteristic wavelengths of the molecules present. The outgoing radiation is processed according to the traditional FTIR spectroscopy method, i.e., performing a Fourier transform operation on the collected signal, thus obtaining the so-called "absorption spectrum," which provides information on the sample's composition. Compared to the traditional FTIR technique, this methodology is particularly useful for analyzing surfaces and solid or liquid samples, including opaque ones or those characterized by high absorption, without complex preparations and with measurement times on the order of a minute.

Finally, the extraction of Extracellular Vesicles (EVs) will be performed from the biological samples of the enrolled patients to characterize the expressed proteins, such as CD147, A33, and FZD10.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Patients undergoing surgery at the U.O.C. of Surgery, with a diagnosis of CRC.
* AIM 2: Subjects without colon disease.
* AIM 3: Subjects with adenoma and high-grade dysplasia.

Exclusion Criteria:

* Subject with any other pathology not included in the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study cohort is comprised of patients with a diagnosis of CRC who underwent surgical intervention, and a cohort of subjects with high-grade dysplasia adenoma, which is considered a precancerous condition.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Variation in serum biomarkers for CRC | From enrollment to the day of the visit after 20 days
  Changes in the concentration of potential serum CRC biomarkers in patients with established CRC pre- and post-surgery, patients with an adenoma with high-grade dysplasia, and subjects with no evidence of disease.

SECONDARY OUTCOMES:
Variation of macroconstituents | From enrollment to the day of the visit after 20 days
  Variation in the macromolecule composition of biological samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Biobank Core Facility, Castellana Grotte, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin-Garcia D, Garcia-Aranda M, Redondo M. Biomarker Identification through Proteomics in Colorectal Cancer. Int J Mol Sci. 2024 Feb 14;25(4):2283. doi: 10.3390/ijms25042283. PMID 38396959
- [Background] Shah SC, Itzkowitz SH. Colorectal Cancer in Inflammatory Bowel Disease: Mechanisms and Management. Gastroenterology. 2022 Mar;162(3):715-730.e3. doi: 10.1053/j.gastro.2021.10.035. Epub 2021 Oct 29. PMID 34757143
- [Background] Sninsky JA, Shore BM, Lupu GV, Crockett SD. Risk Factors for Colorectal Polyps and Cancer. Gastrointest Endosc Clin N Am. 2022 Apr;32(2):195-213. doi: 10.1016/j.giec.2021.12.008. Epub 2022 Feb 22. PMID 35361331